CLINICAL TRIAL: NCT04583891
Title: Evaluating a Mobile Application to Reduce Distress in Breast Cancer Survivors Using an Adaptive Design
Brief Title: Mobile Apps to Reduce Distress in Breast Cancer Survivors Using an Adaptive Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Northwestern University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Philip Chow, Ph.D., Assistant Professor, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 200218; 1R37CA248434-01A1 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-10-12 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Depression, Anxiety; Engagement, Patient
Keywords: Breast Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Patient Participation; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential, Multiple Assignment, Randomized Trial (SMART)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IntelliCare (Experimental): IntelliCare is a self-guided, fully automated suite of apps designed for brief, frequent check-ins to promote skill acquisition. IntelliCare has been shown in both general deployment and human-supported trials to be efficacious in reducing symptoms of depression and anxiety.
  Interventions: Behavioral: IntelliCare; Behavioral: Coaching
- Patient Education (Active Comparator): The patient education app will contain psychoeducational information about distress prevalence and distress management. It will serve as an active control condition to compare with the IntelliCare apps.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: IntelliCare — IntelliCare is a self-guided, fully automated suite of 6 apps designed for brief, frequent check-ins to promote skill acquisition. IntelliCare has been shown in both general deployment and human-supported trials to be efficacious in reducing symptoms of depression and anxiety.
  Arms: IntelliCare
Behavioral: Psychoeducation — The Patient Education app will contain content relevant for general distress management. This includes information about thoughts/worries, prevalence of mood symptoms, CBT strategies for coping with negative affect, and other information typical of education-based mental health apps. The structure of this app will closely mirror patient education websites and apps which mimic the form and structure of apps that target cancer survivors and that primarily provide educational information about cancer and related symptoms.
  Arms: Patient Education
Behavioral: Coaching — The randomization of added coaching vs. no added coaching after 1 week will only be carried out in the IntelliCare group. Coaching is a human supported approach to optimizing the use and benefit of the IntelliCare apps.
  Arms: IntelliCare

SUMMARY:
The overarching goals of this project are to provide the first rigorous test of a scalable and publicly accessible mobile health intervention (IntelliCare) to address emotional distress in women with breast cancer, and to test the impact of human coaching as a way to increase engagement with digital health interventions to improve outcomes. To achieve these goals, an innovative experimental study design, known as a Sequential, Multiple Assignment, Randomized Trial (SMART), will be used to test the effects of the IntelliCare apps on symptoms of depression and anxiety, as well as the added value of human support to improve participant engagement. 313 breast cancer survivors diagnosed within the past 5 years and who screen positive for elevated symptoms of depression and/or anxiety will be recruited. Participants will initially be randomized to receive the IntelliCare apps or app-delivered patient education (control) for 8 weeks, and the impact of the IntelliCare apps on reducing symptoms of depression and anxiety in breast cancer survivors relative to control will be tested (Aim 1). We will monitor the app usage data of participants who receive the IntelliCare apps. Those who are high-engagers will continue to use the apps with no change. Those who are low-to-moderate engagers will be rerandomized after 1 week to either receive added coaching vs. not (i.e., no change) in addition to the apps. The hypothesis is that added coaching to address barriers to app usage will lead to greater engagement with the apps (Aim 2), for low-to-moderate engagers. Finally, semi-structured exit interviews will be conducted with participants that receive the IntelliCare apps and coaching. Interviews will capture survivors' perceptions about the extent to which, and how, tailoring the apps and coaching specifically for breast cancer survivors may improve intervention outcomes and engagement (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years (age 19 if in Nebraska, given age of consent);
2. 0-5 years post-diagnosis of Stage I, II, or III female breast cancer;
3. elevated symptoms of depression as measured by the Patient Health Questionnaire-8 (PHQ-8) score ≥ 10 and/or symptoms of anxiety as measured by the Generalized Anxiety Disorder-7 (GAD-7) score ≥ 8.

Exclusion Criteria:

1. Taking antidepressant medication and have had an appointment to adjust the dosage over the past 2 weeks;
2. mental health condition deemed to interfere with study procedures or put the participant at undue risk based on self-reported history of psychosis or bipolar disorder, or active suicidal ideation that necessitates more intense care;
3. do not have an app-compatible phone (i.e., iOS 10.3 or later or Android 4.0.3 or later);
4. cannot read and speak English (current intervention only available in English).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is not based on self-representation of gender identity.
Enrollment: 313 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants withdrew from the study shortly after being randomized to IntelliCare and never accessed the program. They are therefore not included in any IntelliCare subgroups (i.e., IntelliCare - High Engager, No Coaching; IntelliCare - Low Engager, No Coaching; IntelliCare - Low Engager, Coaching). Subgroup assignment is based on participant engagement with IntelliCare, and because these participants withdrew before engaging with the program, they do not fit into any IntelliCare subgroup.
Groups:
- IntelliCare - High Engager, No Coaching: This arm included participants who received IntelliCare and displayed optimal levels of engagement to the intervention in the first week. These participants were not eligible to receive added coaching after week two. They continued to use IntelliCare as usual.
- IntelliCare - Low Engager, No Coaching: This arm included participants who received IntelliCare and displayed suboptimal levels of engagement to the intervention in the first week. These participants were eligible to receive added coaching after week two. They were randomized to receive no added coaching and continued to use IntelliCare as usual.
- IntelliCare - Low Engager, Coaching: This arm included participants who received IntelliCare and displayed suboptimal levels of engagement to the intervention in the first week. These participants were eligible to receive added coaching after week two. They were randomized to receive added coaching which consisted of an initial phone call with a human coach, a midpoint check-in, and regular messaging with their coach.
Period: Overall Study
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Started | 134 | 38 | 34 | 104
Completed | 130 | 33 | 32 | 94
Not Completed | 4 | 5 | 2 | 10

BASELINE CHARACTERISTICS:
Population: There were 3 enrolled participants who withdrew shortly after being randomized to IntelliCare and never accessed the program. They are not included in any of the IntelliCare subgroups because they were not able to be categorized as high or low engagers.
Groups:
- Total: Total of all reporting groups
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education | Total
Number analyzed (Participants) | 134 | 38 | 34 | 104 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.7) | 50.0 (10.9) | 50.2 (10.9) | 52.2 (10.2) | 51.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 38 | 34 | 104 | 310
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 2 | 5 | 19
  Not Hispanic or Latino | 124 | 36 | 32 | 96 | 288
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 9 | 5 | 4 | 7 | 25
  White | 120 | 32 | 28 | 91 | 271
  More than one race | 2 | 0 | 1 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-8
Description: 8 item scale that measures depression symptoms on a continuous scale. Scores range from 0-24, with a higher score indicating greater severity of symptoms of depression.
Time Frame: Baseline
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 134 | 38 | 34 | 104
score on a scale | 12.1 (4.6) | 11.8 (4.1) | 12.5 (4.5) | 12.7 (4.4)

2. Primary Outcome: Patient Health Questionnaire-8
Description: as for outcome 1
Time Frame: Post 8 weeks
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IntelliCare - High Engager, No Coaching: This arm included participants who received IntelliCare and displayed optimal levels of engagement to the intervention in the first week. These participants were not eligible to receive added coaching after week two. They continued to use IntelliCare as usual.
  Coaching: The randomization of added coaching vs. no added coaching after 1 week will only be carried out in the IntelliCare group. Coaching is a human supported approach to optimizing the use and benefit of the IntelliCare apps.
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 122 | 34 | 32 | 96
score on a scale | 8.1 (5.1) | 10.5 (5.8) | 7.2 (4.4) | 9.4 (4.9)

3. Primary Outcome: Patient Health Questionnaire-8
Description: as for outcome 1
Time Frame: 6 month follow up
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 121 | 32 | 31 | 93
score on a scale | 7.2 (4.9) | 7.4 (4.3) | 7.2 (5.1) | 8.8 (5.5)

4. Primary Outcome: Patient Health Questionnaire-8
Description: as for outcome 1
Time Frame: 12 month follow up
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 120 | 32 | 31 | 90
score on a scale | 6.7 (4.9) | 7.4 (3.9) | 6.6 (5.6) | 8.3 (5.9)

5. Primary Outcome: Generalized Anxiety Disorder-7
Description: 7 item scale that measures anxiety symptoms on a continuous scale. Scores range from 0-21, with a higher score indicating greater severity of symptoms of anxiety.
Time Frame: Baseline
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 134 | 38 | 34 | 104
score on a scale | 11.4 (4.0) | 12.2 (5.0) | 12.4 (5.2) | 12.6 (4.7)

6. Primary Outcome: Generalized Anxiety Disorder-7
Description: as for outcome 5
Time Frame: Post 8 weeks
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 94
score on a scale | 6.9 (4.6) | 7.6 (4.5) | 7.7 (5.1) | 8.9 (5.5)

7. Primary Outcome: Generalized Anxiety Disorder-7
Description: as for outcome 5
Time Frame: 6 month follow up
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 127 | 32 | 30 | 94
score on a scale | 6.3 (5.0) | 7.0 (4.6) | 7.3 (5.7) | 8.0 (5.5)

8. Primary Outcome: Generalized Anxiety Disorder-7
Description: as for outcome 5
Time Frame: 12 month follow up
Population: Breast Cancer Survivors who were classified as high or low engagers and who completed every item of this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 123 | 32 | 32 | 89
score on a scale | 5.7 (5.1) | 6.0 (4.2) | 7.2 (5.6) | 7.5 (5.8)

9. Secondary Outcome: App Engagement From App Sessions
Description: Frequency of unique app sessions from Baseline through 8 weeks based on median number of app sessions
Time Frame: Frequency of unique app sessions from Baseline through 8 weeks
Population: Includes only participants who downloaded their assigned app or intervention.
Measure: Median (Inter-Quartile Range); unit: app sessions
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 134 | 38 | 34 | 102
app sessions
  Week 1 | 12 [8.5 to 15.5] | 6 [3.5 to 8.5] | 7 [5 to 9] | 2 [1 to 3]
  Week 2 | 9 [5 to 13] | 4 [2 to 6] | 4.5 [2 to 7] | 0 [0 to 1]
  Week 3 | 8 [4.5 to 11.5] | 2.5 [1 to 4] | 5 [2.5 to 7.5] | 0 [0 to 0]
  Week 4 | 7 [3.5 to 10.5] | 1 [0 to 4] | 5 [2 to 8] | 0 [0 to 0]
  Week 5 | 6 [3 to 9] | 2 [0.5 to 3.5] | 3.5 [1.5 to 5.5] | 0 [0 to 0]
  Week 6 | 5 [2.5 to 7.5] | 1 [0 to 3] | 4 [2 to 6] | 0 [0 to 0]
  Week 7 | 5 [2 to 8] | 0.5 [0 to 4] | 4.5 [2.5 to 6.5] | 0 [0 to 0]
  Week 8 | 4 [0.5 to 7.5] | 0.5 [0 to 3] | 3.5 [1.5 to 5.5] | 0 [0 to 0]

10. Secondary Outcome: App Engagement From App Session Duration
Description: Duration in seconds of app sessions from Baseline through 8 weeks
Time Frame: Duration in seconds of app sessions from Baseline through 8 weeks
Population: Technical problems led to not being able to extract app engagement based on app session duration from any participants. Data related to the gold standard metric of number of app sessions was captured and reported.
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: App Engagement From App Downloads
Description: Number of apps downloaded from Baseline through 8 weeks
Time Frame: Number of apps downloaded from Baseline through 8 weeks
Population: Technical problems led to not being able to extract app engagement based on number of app downloads from any participants. Data related to the gold standard metric of number of app sessions was captured and reported.
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: 36-Item Short Form Survey - Physical Health
Description: The SF-36 is a 36 item scale that is composed of 2 summary scores that measure health status related to both physical and mental health. Scores for each domain range from 0-100, with higher scores indicating better health status.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 134 | 38 | 34 | 104
score on a scale | 35.5 (40.9) | 41.4 (36.9) | 39.7 (42.2) | 35.7 (39.4)

13. Secondary Outcome: 36-Item Short Form Survey - Physical Health
Description: as for outcome 12
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 129 | 36 | 33 | 98
score on a scale | 44.7 (41.9) | 45.8 (36.6) | 53.8 (41.5) | 44.5 (40.2)

14. Secondary Outcome: 36-Item Short Form Survey - Physical Health
Description: as for outcome 12
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 127 | 33 | 31 | 96
score on a scale | 60.3 (42.1) | 51.5 (41.0) | 56.5 (45.2) | 49.0 (40.1)

15. Secondary Outcome: 36-Item Short Form Survey - Physical Health
Description: as for outcome 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 92
score on a scale | 65.9 (41.3) | 52.3 (41.6) | 56.0 (42.5) | 56.8 (41.8)

16. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 12
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 134 | 38 | 34 | 104
score on a scale | 54.2 (16.3) | 47.9 (16.8) | 48.2 (14.6) | 48.6 (16.9)

17. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 12
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 129 | 36 | 33 | 98
score on a scale | 62.7 (17.5) | 59.3 (18.2) | 57.8 (19.5) | 55.3 (18.3)

18. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 12
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 33 | 30 | 96
score on a scale | 69.6 (16.4) | 60.7 (19.0) | 60.3 (20.9) | 61.3 (17.4)

19. Secondary Outcome: 36-Item Short Form Survey - Mental Health
Description: as for outcome 12
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 92
score on a scale | 68.7 (16.9) | 66.2 (14.6) | 64.5 (18.7) | 63.1 (19.6)

20. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form
Description: Fatigue will be measured using the MFSI-SF, which is a 30 item self-report measure comprised of five subscales (general, emotional, physical, mental, vigor) and a total fatigue score. Each subscale score ranges from 0 to 24. The Total MSFI-SF score is calculated by adding the general, physical, emotional and mental subscale scores and subtracting vigor subscale score. Total MFSI-SF score ranges from 0 to 96 with a higher score indicating higher levels of cancer-related fatigue experienced by the patient.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 35 | 32 | 95
score on a scale | 35.4 (19.5) | 38.8 (16.4) | 42.9 (17.4) | 42.0 (19.8)

21. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form
Description: as for outcome 20
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 120 | 35 | 30 | 88
score on a scale | 25.3 (20.1) | 29.5 (19.3) | 27.2 (20.1) | 31.3 (22.5)

22. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form
Description: as for outcome 20
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 118 | 30 | 25 | 87
score on a scale | 21.1 (21.1) | 26.8 (19.2) | 24.6 (19.4) | 29.5 (24.3)

23. Secondary Outcome: Multidimensional Fatigue Symptom Inventory-Short Form
Description: as for outcome 20
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 117 | 33 | 31 | 85
score on a scale | 19.7 (22.7) | 24.0 (18.1) | 20.5 (22.2) | 25.8 (23.2)

24. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index contains 19 self-rated questions that assesses sleep quality and disturbances. Global scores range from 0-21, with a score of 5 or more indicating poor sleep quality. The higher the score, the worse the sleep quality.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 123 | 31 | 31 | 100
score on a scale | 10.7 (4.1) | 10.8 (3.5) | 10.2 (4.0) | 11.1 (4.3)

25. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: as for outcome 24
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 118 | 31 | 30 | 85
score on a scale | 9.8 (4.0) | 9.3 (3.4) | 8.5 (4.2) | 9.9 (4.3)

26. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: as for outcome 24
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 112 | 30 | 28 | 84
score on a scale | 8.9 (3.8) | 10.1 (3.5) | 8.5 (4.0) | 9.8 (4.6)

27. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: as for outcome 24
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 110 | 30 | 31 | 80
score on a scale | 8.7 (4.0) | 9.6 (3.6) | 8.0 (3.5) | 9.5 (4.2)

28. Secondary Outcome: Alcohol Use Disorders Identification Test
Description: The Alcohol Use Disorders Identification Test contains 10 questions (each question is scored 0-4). The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 132 | 36 | 34 | 101
score on a scale | 2.3 (3.4) | 4.0 (5.4) | 2.2 (2.9) | 1.7 (2.8)

29. Secondary Outcome: Alcohol Use Disorders Identification Test
Description: as for outcome 28
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 36 | 33 | 98
score on a scale | 2.0 (3.4) | 3.5 (5.1) | 1.9 (2.6) | 1.5 (2.7)

30. Secondary Outcome: Alcohol Use Disorders Identification Test
Description: as for outcome 28
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 32 | 29 | 95
score on a scale | 1.7 (2.9) | 3.3 (5.3) | 1.6 (2.6) | 1.5 (2.6)

31. Secondary Outcome: Alcohol Use Disorders Identification Test
Description: as for outcome 28
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 32 | 31 | 91
score on a scale | 2.0 (3.2) | 3.7 (5.9) | 1.7 (3.0) | 1.7 (3.1)

32. Secondary Outcome: PROMIS Global Mental Health v1.2
Description: The PROMIS Global Mental Health scale v1.2 contains 4 items that measure mental health. Each question is scored on a 1-5 scale with a raw score total range of 4-20. The raw scores are then transformed into a T-score where higher scores indicate better overall health. PROMIS uses T-scores to standardize results, with a mean of 50 and a standard deviation (SD) of 10 for the general U.S. population. A higher T-score for mental health indicates a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 131 | 37 | 34 | 101
T-score | 39.5 (6.3) | 38.8 (6.1) | 37.6 (5.6) | 38.4 (7.0)

33. Secondary Outcome: PROMIS Global Mental Health v1.2
Description: as for outcome 32
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 36 | 32 | 95
T-score | 42.6 (7.1) | 41.5 (6.0) | 42.4 (5.6) | 40.3 (7.0)

34. Secondary Outcome: PROMIS Global Mental Health v1.2
Description: as for outcome 32
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 30 | 96
T-score | 45.2 (8.6) | 43.7 (6.6) | 43.0 (6.6) | 41.4 (7.9)

35. Secondary Outcome: PROMIS Global Mental Health v1.2
Description: as for outcome 32
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 91
T-score | 45.5 (8.5) | 45.2 (6.0) | 44.8 (6.6) | 42.6 (8.3)

36. Secondary Outcome: PROMIS Satisfaction With Sex Life
Description: The PROMIS Satisfaction with Sex Life scale v.20 contains 5 items that measure satisfaction with one's sex life. Each question is scored on a 1-5 scale with a total score range of 5-25. Higher scores indicate higher satisfaction with one's sex life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 127 | 35 | 34 | 101
score on a scale | 9.4 (5.0) | 8.9 (4.6) | 10.6 (6.5) | 9.2 (5.0)

37. Secondary Outcome: PROMIS Satisfaction With Sex Life
Description: as for outcome 36
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 119 | 35 | 31 | 95
score on a scale | 9.3 (5.1) | 9.1 (5.1) | 11.7 (6.3) | 9.9 (5.1)

38. Secondary Outcome: PROMIS Satisfaction With Sex Life
Description: as for outcome 36
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 123 | 32 | 30 | 95
score on a scale | 10.5 (5.9) | 9.7 (5.6) | 11.6 (5.9) | 10.2 (5.7)

39. Secondary Outcome: PROMIS Satisfaction With Sex Life
Description: as for outcome 36
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 121 | 33 | 30 | 90
score on a scale | 10.6 (6.1) | 10.4 (6.0) | 12.0 (6.5) | 10.5 (5.9)

40. Secondary Outcome: UAMS Health Literacy Measure
Description: The UAMS Health Literacy measure consists of 3 items that assess health literacy. Each question is scored on a 1-5 scale, with a possible total score range of 3-15. Higher scores indicate worse health literacy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 133 | 38 | 34 | 104
score on a scale | 10.3 (1.2) | 10.7 (1.0) | 10.3 (1.3) | 10.4 (1.1)

41. Secondary Outcome: UAMS Health Literacy Measure
Description: as for outcome 40
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 36 | 31 | 98
score on a scale | 10.5 (1.1) | 10.4 (1.3) | 10.0 (1.7) | 10.5 (1.2)

42. Secondary Outcome: UAMS Health Literacy Measure
Description: as for outcome 40
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 127 | 32 | 30 | 96
score on a scale | 10.5 (1.1) | 10.7 (1.0) | 10.7 (0.8) | 10.7 (1.2)

43. Secondary Outcome: UAMS Health Literacy Measure
Description: as for outcome 40
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 32 | 32 | 92
score on a scale | 10.6 (1.1) | 10.6 (0.8) | 10.4 (1.2) | 10.7 (0.9)

44. Secondary Outcome: Penn State Worry Questionnaire
Description: The Penn State Worry Questionnaire consists of 16 items that assess the trait of worry. Each question is scored on a 1-5 scale with a possible total score range of 16-80. Higher scores indicate higher levels of trait worry.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 124 | 36 | 32 | 97
score on a scale | 56.8 (12.7) | 57.8 (13.7) | 61.3 (14.1) | 59.5 (12.7)

45. Secondary Outcome: Penn State Worry Questionnaire
Description: as for outcome 44
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 120 | 34 | 30 | 91
score on a scale | 53.1 (12.9) | 54.0 (12.8) | 54.2 (14.3) | 55.0 (12.4)

46. Secondary Outcome: Penn State Worry Questionnaire
Description: as for outcome 44
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 122 | 32 | 27 | 91
score on a scale | 50.1 (13.9) | 50.8 (10.2) | 55.9 (15.5) | 55.0 (13.5)

47. Secondary Outcome: Penn State Worry Questionnaire
Description: as for outcome 44
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 118 | 32 | 31 | 91
score on a scale | 48.8 (13.0) | 49.4 (12.3) | 51.9 (14.6) | 54.4 (14.4)

48. Secondary Outcome: Ten Item Personality Inventory- Extraversion
Description: The Ten Item Personality Inventory consists of 10 items that assess the Big 5 personality domains (i.e., conscientiousness, openness, agreeableness, extraversion, neuroticism). Extraversion is assessed by 2 items, each of which is scored on a 1-7 scale and the responses are summed for a total Extraversion score. Therefore, scores for Extraversion range from 2-14. Higher scores indicates higher levels of Extraversion.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 134 | 38 | 34 | 100
score on a scale | 8.0 (3.5) | 8.1 (3.5) | 8.8 (3.7) | 7.4 (3.3)

49. Secondary Outcome: Ten Item Personality Inventory - Extraversion
Description: as for outcome 48
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 36 | 32 | 98
score on a scale | 8.1 (3.2) | 8.2 (3.4) | 8.7 (3.9) | 7.3 (3.3)

50. Secondary Outcome: Ten Item Personality Inventory - Extraversion
Description: as for outcome 48
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 32 | 30 | 95
score on a scale | 8.2 (3.3) | 8.1 (3.3) | 8.4 (3.2) | 7.8 (3.1)

51. Secondary Outcome: Ten Item Personality Inventory - Extraversion
Description: as for outcome 48
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 91
score on a scale | 8.3 (3.1) | 7.9 (3.2) | 8.8 (3.5) | 8.0 (3.3)

52. Secondary Outcome: Ten Item Personality Inventory - Agreeableness
Description: The Ten Item Personality Inventory consists of 10 items that assess the Big 5 personality domains (i.e., conscientiousness, openness, agreeableness, extraversion, neuroticism). Agreeableness is assessed by 2 of the items, each of which is scored on a 1-7 scale and the responses are summed for a total Agreeableness score. Therefore, scores for Agreeableness range from 2-14. Higher scores indicates higher levels of Agreeableness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 133 | 38 | 34 | 101
score on a scale | 10.9 (2.2) | 10.2 (2.3) | 10.3 (2.0) | 10.2 (2.6)

53. Secondary Outcome: Ten Item Personality Inventory - Agreeableness
Description: as for outcome 52
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 129 | 36 | 32 | 98
score on a scale | 11.1 (2.3) | 10.9 (2.3) | 11.0 (2.4) | 10.7 (2.6)

54. Secondary Outcome: Ten Item Personality Inventory - Agreeableness
Description: as for outcome 52
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 127 | 32 | 29 | 96
score on a scale | 11.2 (2.3) | 10.8 (2.2) | 11.1 (2.1) | 10.7 (2.5)

55. Secondary Outcome: Ten Item Personality Inventory - Agreeableness
Description: as for outcome 52
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 91
score on a scale | 11.2 (2.5) | 10.7 (2.2) | 10.6 (2.3) | 11.0 (2.3)

56. Secondary Outcome: Ten Item Personality Inventory - Conscientiousness
Description: The Ten Item Personality Inventory consists of 10 items that assess the Big 5 personality domains (i.e., conscientiousness, openness, agreeableness, extraversion, neuroticism). Conscientiousness is assessed by 2 of the items, each of which is scored on a 1-7 scale and the responses are summed for a total Conscientiousness score. Therefore, scores for Conscientiousness range from 2-14. Higher scores indicates higher levels of Conscientiousness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 132 | 38 | 34 | 102
score on a scale | 11.0 (2.6) | 10.8 (2.6) | 10.5 (2.6) | 10.9 (2.6)

57. Secondary Outcome: Ten Item Personality Inventory - Conscientiousness
Description: as for outcome 56
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 36 | 31 | 98
score on a scale | 11.2 (2.2) | 10.4 (3.0) | 11.0 (2.8) | 10.7 (2.7)

58. Secondary Outcome: Ten Item Personality Inventory - Conscientiousness
Description: as for outcome 56
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 32 | 30 | 96
score on a scale | 11.3 (2.5) | 10.8 (2.7) | 10.9 (2.7) | 10.7 (2.7)

59. Secondary Outcome: Ten Item Personality Inventory - Conscientiousness
Description: as for outcome 56
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 33 | 32 | 88
score on a scale | 11.2 (2.4) | 11.0 (2.7) | 10.0 (2.8) | 11.1 (2.5)

60. Secondary Outcome: Ten Item Personality Inventory - Neuroticism
Description: The Ten Item Personality Inventory consists of 10 items that assess the Big 5 personality domains (i.e., conscientiousness, openness, agreeableness, extraversion, neuroticism). Neuroticism is assessed by 2 of the items, each of which is scored on a 1-7 scale and the responses are summed for a total Neuroticism score. Therefore, scores for Neuroticism range from 2-14. Higher scores indicates higher levels of Neuroticism.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 132 | 38 | 33 | 103
score on a scale | 7.6 (2.7) | 7.7 (2.6) | 6.6 (2.7) | 7.3 (2.8)

61. Secondary Outcome: Ten Item Personality Inventory - Neuroticism
Description: as for outcome 60
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 35 | 32 | 97
score on a scale | 8.5 (2.7) | 8.5 (2.5) | 8.3 (2.8) | 7.9 (2.8)

62. Secondary Outcome: Ten Item Personality Inventory - Neuroticism
Description: as for outcome 60
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 33 | 30 | 96
score on a scale | 8.9 (3.0) | 8.5 (2.5) | 8.4 (2.5) | 8.2 (2.8)

63. Secondary Outcome: Ten Item Personality Inventory - Neuroticism
Description: as for outcome 60
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 125 | 33 | 32 | 91
score on a scale | 9.5 (2.7) | 8.9 (2.6) | 8.3 (2.8) | 8.4 (2.9)

64. Secondary Outcome: Ten Item Personality Inventory - Openness
Description: The Ten Item Personality Inventory consists of 10 items that assess the Big 5 personality domains (i.e., conscientiousness, openness, agreeableness, extraversion, neuroticism). Openness is assessed by 2 of the items, each of which is scored on a 1-7 scale and the responses are summed for a total Openness score. Therefore, scores for Openness range from 2-14. Higher scores indicates higher levels of Openness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 133 | 38 | 34 | 102
score on a scale | 10.1 (2.5) | 9.7 (2.3) | 10.8 (2.0) | 9.6 (2.5)

65. Secondary Outcome: Ten Item Personality Inventory - Openness
Description: as for outcome 64
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 128 | 36 | 32 | 98
score on a scale | 10.2 (2.3) | 10.2 (2.5) | 10.5 (2.0) | 9.6 (2.7)

66. Secondary Outcome: Ten Item Personality Inventory - Openness
Description: as for outcome 64
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 30 | 96
score on a scale | 10.2 (2.5) | 10.6 (2.7) | 10.5 (2.1) | 10.2 (2.3)

67. Secondary Outcome: Ten Item Personality Inventory - Openness
Description: as for outcome 64
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 126 | 33 | 32 | 90
score on a scale | 10.4 (2.4) | 10.0 (2.6) | 10.2 (2.5) | 10.2 (2.7)

68. Secondary Outcome: TWente Engagement With Ehealth Technologies Scale (TWEETS)
Description: The TWEETS scale consists of 9 items on a 5-point Likert scale (0-4). Of the 9 items, 3 are aimed at assessing behavioral engagement, 3 on cognitive engagement, and 3 of affective engagement. Higher scores indicate higher levels on each of the engagement domains.
Time Frame: Baseline
Population: This measure was not administered because it was deemed to be redundant with the other intervention engagement and adherence measures. It was omitted to reduce participant burden.
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

69. Secondary Outcome: TWente Engagement With Ehealth Technologies Scale (TWEETS)
Description: as for outcome 68
Time Frame: 8 weeks
Population: as for outcome 68
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

70. Secondary Outcome: TWente Engagement With Ehealth Technologies Scale (TWEETS)
Description: as for outcome 68
Time Frame: 6 months
Population: as for outcome 68
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

71. Secondary Outcome: TWente Engagement With Ehealth Technologies Scale (TWEETS)
Description: as for outcome 68
Time Frame: 12 months
Population: as for outcome 68
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

72. Other Pre Specified Outcome: Digital Intervention Evaluation Questionnaire
Description: A 12-item questionnaire with subscales of perceived utility and perceived impact of digital interventions. Each item is rated on a 0 (not at all) to 5 (very) scale and the items are summed to compute a total score ranging from 0-60. Higher scores indicate higher perceived utility and impact of a digital intervention.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 132 | 36 | 33 | 100
score on a scale | 27.8 (10.5) | 25.7 (10.4) | 30.4 (9.7) | 23.5 (10.7)

73. Other Pre Specified Outcome: Digital Intervention Adherence Questionnaire
Description: A 26 item questionnaire that assesses perceived adherence to a digital intervention due to barriers to use. Each item is scored on a 0 (not at all) to 2 (very) scale and the items are summed to compute a total score ranging from 0-52. Higher scores indicate lower perceived adherence to a digital intervention due to barriers to use.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 132 | 36 | 33 | 100
score on a scale | 7.6 (7.1) | 10.6 (9.3) | 7.3 (6.0) | 5.1 (5.9)

74. Post Hoc Outcome: Limited List of Questions for Exit Interview
Description: The purpose of collecting this data was to explore how the intervention could be improved upon in future trials. Only those that receive the IntelliCare apps will be administered a qualitative interview that contains items assessing how the app intervention met their needs as a breast cancer survivor and possible changes to improve fit. Study staff will administer this interview on the phone and manually type in the participant responses during the interview. 10 questions will assess overall impressions of the IntelliCare app program to inform how it could be improved upon for future trials. When new data no longer adds new information or a new theme to the analysis, the theme is considered sufficiently explored and important. A numerical threshold for theme importance in qualitative analysis is not important, as this can lead to losing valuable, nuanced insights.
Time Frame: 8 weeks
Population: The data collected were qualitative based on interviews with participants who received IntelliCare. The "Patient Education" participants did not receive the Intellicare App. The count of participants that endorsed each theme is provided, however, it is important to stress that the goal was to identify meaningful patterns and concepts within the data, not just count how many people mention a theme.
Measure: Count of Participants; unit: Participants
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
Number analyzed (Participants) | 44 | 23 | 19 | 0
Participants
  More variety of activities in the behavioral activation portion of the intervention | 3 | 4 | 4 | 0
  Make loading pictures easier | 2 | 3 | 3 | 0
  Create a progress report for users as they use the app over time | 4 | 1 | 0 | 0
  Include cancer related examples in the activities in the app to make them more relatable | 17 | 8 | 9 | 0
  Have a way for users to connect with one another directly to provide emotional support | 8 | 1 | 0 | 0
  Want more variety of activities and exercises to choose from to learn additional skills | 10 | 6 | 3 | 0

ADVERSE EVENTS:
Time Frame: through study completion, up to 1 year
Description: Adverse Event: an undesirable and unintended result of therapy, intervention or interaction experienced by a subject participating in a research study.
Arm/Group | IntelliCare - High Engager, No Coaching | IntelliCare - Low Engager, No Coaching | IntelliCare - Low Engager, Coaching | Patient Education
All-Cause Mortality (participants affected / at risk) | 1/137 | 0/38 | 0/34 | 2/104
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/38 | 0/34 | 0/104
Other Adverse Events (participants affected / at risk) | 0/137 | 0/38 | 0/34 | 0/104

LIMITATIONS AND CAVEATS:
Technical problems led to not being able to extract app engagement based on app session duration and number of app downloads from any participants. The TWente Engagement With Ehealth Technologies Scale (TWEETS) was not administered as it was redundant with the other intervention evaluation and adherence measures. These have been recorded in the Results by including "0" participants analyzed and providing an explanation in the Analysis Population Description for why data cannot be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04583891/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04583891/SAP_001.pdf
  • Informed Consent Form (2021-07-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04583891/ICF_002.pdf